CLINICAL TRIAL: NCT06431906
Title: TRANSDERMAL FENTANYL AS A FORM OF REBOUND PAIN REDUCTION IN FAST TRACK PROGRAMME IN PRIMARY KNEE ARTHROPLASTY. Prospective Observational Non-inferiority Study Versus Morphine PCA.
Brief Title: Transdermal Fentanyl as a Form of Rebound Pain Reduction in Fast Track Programme in Primary Knee Arthroplasty.
Acronym: FENTRA
Status: Not yet recruiting | Type: Observational
Sponsor: Oscar Diaz-Cambronero (Other)
Responsible Party: Sponsor-Investigator, Oscar Diaz-Cambronero, MÉDICO ADJUNTO ANESTESIOLOGÍA, Hospital Universitario La Fe
Organization: Hospital Universitario La Fe (Other)
Other Study IDs: FEN
Record Dates: First submitted 2024-04-30; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
Keywords: fentanyl; morphine PCA; rebound pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- transdermal fentanyl: Subjects receiving a transdermal fentanyl patch for postoperative pain control will be included here.
- morphine PCA: Subjects receiving a morphine PCA for postoperative pain control will be included here.

SUMMARY:
Total knee arthroplasty is a common surgery in routine clinical practice that, although it achieves an improvement in the functionality and quality of life of patients, it causes intense postoperative pain. In this regard, locoregional block techniques are commonly used for the immediate postoperative period. However, these techniques have the disadvantage of being of limited duration and the appearance of so-called "rebound pain" when their effect wears off. To counteract this problem and maintain adequate analgesic control over a longer period of time, the use of a transdermal fentanyl patch seems to be a good option, with advantages over the traditional approach of placing a morphine PCA.

Specifically, the aims of the study are: the evaluation of the decrease in the rate of rebound pain after locoregional techniques using a transdermal fentanyl patch after primary knee arthroplasty, as well as the evaluation of non-inferiority in terms of functional recovery, analgesic efficacy and adverse effects compared to morphine PCA.

Methods: This will be a prospective observational cohort study, with a total N of 106 patients undergoing total knee arthroplasty who meet the study inclusion criteria. The numerical pain rating scale score will be collected at 6,8,12,24 and 26h from which the "rebound pain score" will be calculated. The need for pharmacological rescue will be assessed as well as the appearance of adverse effects at 12, 24 and 36h and finally the QoR15 scale will be assessed at 36h.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA from now on) is a frequent surgery in routine clinical practice in constant evolution and improvement, with the objective being the earliest possible functional recovery of these patients, the role of the anaesthesiologist being fundamental in this sense throughout the perioperative period since, as we know, it is a surgery that improves the mobility and quality of life of the patient, but causes intense postoperative pain during the first 24 to 72 hours, it is a surgery that improves the patient's mobility and quality of life, but causes intense postoperative pain during the first 24 to 72 hours, a very important factor to take into account in these patients since it is known that adequate postoperative pain control promotes ambulation and the possibility of physiotherapy for the patient, This leads to an early recovery, a lower rate of complications (such as deep vein thrombosis or nosocomial infection) and a shorter hospital stay, allowing the strategy known as "fast-track" to be carried out, which would consist of achieving functional recovery and discharge as early as possible, this being the current trend in management by most trauma teams dedicated to this field, since it results in a decrease in morbidity and greater patient satisfaction. In relation to this approach, as has been mentioned, multiple studies have shown that one of the main causes of delayed hospital discharge is poor pain control and mobilisation problems.

Therefore, adequate postoperative pain control will be important in this surgery. This control could be achieved with a combination of locoregional techniques such as peripheral nerve blocks of the adductor canal (BCA) and the so-called "Infiltration between the Popliteal Artery and the Capsule of the Knee" (IPACK) together with conventional analgesia such as NSAIDs, paracetamol, metamizole and, if this is not sufficient, opioids.

The locoregional techniques mentioned (BCA + IPACK) have demonstrated their efficacy in controlling immediate postoperative pain in this type of surgery in multiple studies. The first of these, BCA, provides analgesia in the anteromedial area of the knee, avoiding the femoral nerve block with the consequent weakness of the quadriceps. The second of these, IPACK, is a relatively novel technique described to achieve analgesia in the posterior capsule of the knee that is achieved by blocking the popliteal plexus formed by the articular sensory branches of the tibial and obturator nerves arranged around the popliteal artery and vein without involving the motor branches of the tibial and peroneal nerves, avoiding the motor block resulting from performing a block of the sciatic nerve at the popliteal level.

From all of the above, we can deduce that both techniques are effective individually, but even more so, as is logical, in combination, allowing the entire joint territory to be covered with the least possible impairment of motor function, which will be of particular relevance in terms of starting the patient's mobilisation earlier, which is definitely an advantage over traditional femoral and sciatic nerve block techniques.

However, the duration of nerve blocks is less than 24h, which is a problem, since the period of maximum incidence of postoperative pain has not yet been completed and it is possible that just at this time (12-24h after the block, when the effect of the block ends) what is known as "rebound pain" may appear, considered a possible adverse effect of peripheral nerve blocks that is becoming increasingly important, as studies dedicated to its study emerge.

There are multiple definitions of rebound pain in the literature, but objectively, we can say that it is a quantifiable difference between scores on pain scales when the block works and when it stops working. Its incidence is not well established, although some studies report that it appears in up to 40% of cases receiving some type of peripheral nerve block, although its incidence in the type of patient on whom this study is to be performed has not been specifically defined in the literature available to date. As for its characteristics, we can say that it appears suddenly at 12-24h, lasting 3-6h, described by many patients as a burning sensation that worsens at night. Logically, this will have a negative impact on the patient's recovery, and will require the use of rescue drugs, mainly intravenous opioids.

To date, the pathophysiological mechanisms by which it occurs continue to be the subject of debate. It is definitely a sum of mechanical and chemical factors (neurotoxicity of local anaesthetics, hyperactivity of nerve fibres, hyperexcitability of nociceptors, direct mechanical damage, etc.) in patients with predisposing factors (young people, women, orthopaedic surgery, pre-existing pain, etc.).

Once its existence is known, the two most important aspects will be its proper diagnosis and definition, on the one hand, and its prevention and treatment, on the other.

In terms of its detection, rebound pain will be diagnosed when a difference in pain scale scores is observed at the end of the peripheral blockade effect, which is usually 12-24 hours after it has been performed. To quantify it, most studies use serial scores on the numerical pain scale (NRS), and even the "rebound pain score" has been described, which is obtained by subtracting the lowest pain score in the first 12 hours before the end of the block action from the highest pain score in the first 12 hours after the end of the block action.

In prevention and treatment, a multifactorial approach will be essential, employing pharmacological and non-pharmacological strategies (mainly patient education). Among the pharmacological strategies, there are multiple strategies that have been shown to reduce the rate of rebound pain but among which there is no clear consensus: the use of adjuvants such as dexamethasone or alpha2-agonists, which not only prolong the duration of the block but also seem to exert a neuromodulatory effect; use of continuous infusion catheters instead of a single puncture; combination of various types of peripheral blockade or intra-articular infiltration. Another option, this one highly recommended in general, is the initiation of analgesic treatment prior to the end of the blockade effect, since once it occurs, it will be very difficult to control, making it necessary to rescue with intravenous drugs, mainly major opioids such as morphine in the form of a PCA pump, an analgesic modality that has demonstrated its effectiveness but which has a number of negative aspects such as: the need for personnel capable of handling the device and a learning process on the part of the patient; the possibility of programming and medication administration errors; an increase in economic cost; in addition to the consequent limitation of mobility derived from the connection to the PCA device or the delay in discharge due to the patient being under intravenous treatment.

However, a new possibility has emerged in the form of the transdermal fentanyl patch (TFP); a skin patch that constantly releases fentanyl into the bloodstream according to the dose applied, traditionally used in the control of chronic pain but whose efficacy has already been demonstrated in multiple types of surgery such as abdominal, urological and orthopaedic procedures such as hip and knee surgery. Fentanyl is a major opioid with 75-100 times the potency of morphine. Because it is highly lipid soluble and has a low molecular weight (337da), it is ideal for administration in this transdermal format; it also produces fewer cardiovascular effects than other opioids and has a lower risk of histamine release than morphine. Once applied, the patch has a slow onset of action with a plasma peak in about 12-15h and stable plasma concentrations thereafter for approximately 72h of duration. It has many advantages over other forms of analgesia, such as ease of administration, reduced possibility of dosing error, no need for venous access, low risk of infection and easier to obtain than devices such as the PCA pump.

The main drawback to its use as a form of postoperative analgesia lies in its slow onset of action, since, as mentioned, its plasma peak would be reached at 15h, which makes it unsuitable for acute pain control. However, if applied at the time of surgery, it could superimpose its analgesia on the end of the analgesic effect of the peripheral nerve block, thus avoiding the appearance of rebound pain or at least reducing its rate of appearance.

Therefore, several positive aspects could be derived from this alternative: convenience in its dosage, reduction of resources necessary for the adequate control and functioning of a morphine PCA and improvement in postoperative pain control, resulting in an increase in the degree of patient satisfaction and autonomy and a shorter hospital stay.

With all of the above, we propose the hypothesis that the transdermal fentanyl patch is an effective postoperative analgesic strategy in primary knee arthroplasty after the disappearance of the analgesic effect of the peripheral nerve blocks Canal of the Adductors + IPACK, achieving a decrease in the rate of "rebound pain", our main objective being therefore the following:

Main objective:

- To evaluate the decrease in the rate of rebound pain after primary knee arthroplasty with the use of transdermal fentanyl patch versus morphine PCA.

To do all this we will use objective and validated tools. For the measurement of the first objective we will use the "Rebound Pain Score", described above.

As for the secondary objectives that we propose to evaluate in this work, on the one hand, we want to focus on assessing the functional recovery of patients, for which we will use the QoR 15 scale, developed from the QoR40 (27), which has proven to be a suitable tool for measuring postoperative recovery (28); and on the other hand, to compare the two pharmacological modalities under study in terms of analgesic quality and adverse effects. Therefore, the following would be our secondary objectives:

Secondary objectives:

* To assess the non-inferiority in terms of functional recovery after primary knee arthroplasty of the transdermal fentanyl patch versus morphine PCA.
* To assess the analgesic non-inferiority in terms of postoperative analgesia after primary knee arthroplasty of the 25mcg/h transdermal fentanyl patch versus morphine PCA.
* To assess the non-inferiority in terms of incidence of adverse effects in postoperative total knee arthroplasty of 25mcg/h transdermal fentanyl patch versus morphine PCA.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary knee arthroplasty ASA I-III between 18 and 80 years of age who have received a transdermal fentanyl patch or morphine PCA as part of their postoperative analgesic strategy

Exclusion Criteria:

* Prior opioid treatment.
* History of previous opioid adverse effects.
* History of PONV.
* History of medical history that conditions baseline alteration of the data to be collected.
* Contraindication to neuroaxial techniques.
* Difficulty in understanding the scales used.
* Patient's refusal.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing primary knee arthroplasty ASA I-III between 18 and 80 years of age who have received a transdermal fentanyl patch or morphine PCA as part of their postoperative analgesic strategy.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
- Responders to the decrease in the rate of "rebound pain" with the use of transdermal fentanyl patch relative to morphine PCA: | 6,8,12,24 and 36hours after the lock
  - Rebound pain score (RPS): Defined as the result of subtracting the minimum score on the pain scale the first 12 hours before the end of action of the peripheral blockade from the maximum score on the pain scale the first 12 hours after the disappearance of the action of the peripheral blockade. To calculate this variable, the numerical pain scale score will be collected 6, 8, 12, 24 and 36 hours after the peripheral nerve block.

SECONDARY OUTCOMES:
non-inferiority of PFT vs PCA morphine in terms of early postoperative recovery: | 48 hours in the postoperative period
  Quality of post-surgical recovery using the QoR 15 scale at 48 hours
non-inferiority of PFT vs. morphine PCA in terms of post-surgical analgesia: | 48 hours in the postoperative period
  * Need for prescribed pharmacological rescue at 12 hours: Yes or no
  * Need for pharmacological rescue at 24 hours: Yes or no
  * Need for pharmacological rescue at 48 hours: Yes or No
non-inferiority of PFT vs morphine PCA in terms of adverse effects: | 48 hours in the postoperative period
  Presence or not of the following adverse effects at 48 hours: pruritus, urinary retention/bladder catheterisation, constipation or abdominal distention, limited mobility, tremor.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sathitkarnmanee T, Tribuddharat S, Noiphitak K, Theerapongpakdee S, Pongjanyakul S, Huntula Y, Thananun M. Transdermal fentanyl patch for postoperative analgesia in total knee arthroplasty: a randomized double-blind controlled trial. J Pain Res. 2014 Aug 1;7:449-54. doi: 10.2147/JPR.S66741. eCollection 2014. PMID 25120375
- [Background] Matsumoto S, Matsumoto K, Iida H. Transdermal fentanyl patch improves post-operative pain relief and promotes early functional recovery in patients undergoing primary total knee arthroplasty: a prospective, randomised, controlled trial. Arch Orthop Trauma Surg. 2015 Sep;135(9):1291-7. doi: 10.1007/s00402-015-2265-z. Epub 2015 Jun 26. PMID 26112273
- [Background] Hall MJ, Dixon SM, Bracey M, MacIntyre P, Powell RJ, Toms AD. A randomized controlled trial of postoperative analgesia following total knee replacement: transdermal Fentanyl patches versus patient controlled analgesia (PCA). Eur J Orthop Surg Traumatol. 2015 Aug;25(6):1073-9. doi: 10.1007/s00590-015-1621-6. Epub 2015 Mar 11. PMID 25753087
- [Background] Kehlet H, Thienpont E. Fast-track knee arthroplasty -- status and future challenges. Knee. 2013 Sep;20 Suppl 1:S29-33. doi: 10.1016/S0968-0160(13)70006-1. PMID 24034592
- [Background] Lindberg-Larsen M, Petersen PB, Corap Y, Gromov K, Jorgensen CC, Kehlet H; Centre for Fast-track Hip and Knee Replacement Collaborating Group. Fast-track revision hip arthroplasty: a multicenter cohort study on 1,345 elective aseptic major component revision hip arthroplasties. Acta Orthop. 2022 Feb 23;93:341-347. doi: 10.2340/17453674.2022.2196. PMID 35195270
- [Background] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648
- [Background] Abdullah MA, Abu Elyazed MM, Mostafa SF. The Interspace Between Popliteal Artery and Posterior Capsule of the Knee (IPACK) Block in Knee Arthroplasty: A Prospective Randomized Trial. Pain Physician. 2022 May;25(3):E427-E433. PMID 35652772
- [Background] Tang X, Jiang X, Lei L, Zhu W, Fu Z, Wang D, Chen J, Ning N, Zhou Z. IPACK (Interspace between the Popliteal Artery and the Capsule of the Posterior Knee) Block Combined with SACB (Single Adductor Canal Block) Versus SACB for Analgesia after Total Knee Arthroplasty. Orthop Surg. 2022 Nov;14(11):2809-2821. doi: 10.1111/os.13263. Epub 2022 Sep 20. PMID 36125191
- [Background] Ochroch J, Qi V, Badiola I, Grosh T, Cai L, Graff V, Nelson C, Israelite C, Elkassabany NM. Analgesic efficacy of adding the IPACK block to a multimodal analgesia protocol for primary total knee arthroplasty. Reg Anesth Pain Med. 2020 Oct;45(10):799-804. doi: 10.1136/rapm-2020-101558. Epub 2020 Aug 31. PMID 32868483
- [Background] Kampitak W, Tanavalee A, Ngarmukos S, Tantavisut S. Motor-sparing effect of iPACK (interspace between the popliteal artery and capsule of the posterior knee) block versus tibial nerve block after total knee arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2020 Apr;45(4):267-276. doi: 10.1136/rapm-2019-100895. Epub 2020 Feb 4. PMID 32024676
- [Background] Guo J, Hou M, Shi G, Bai N, Huo M. iPACK block (local anesthetic infiltration of the interspace between the popliteal artery and the posterior knee capsule) added to the adductor canal blocks versus the adductor canal blocks in the pain management after total knee arthroplasty: a systematic review and meta-analysis. J Orthop Surg Res. 2022 Aug 12;17(1):387. doi: 10.1186/s13018-022-03272-5. PMID 35962410
- [Background] Zheng FY, Liu YB, Huang H, Xu S, Ma XJ, Liu YZ, Chu HC. The impact of IPACK combined with adductor canal block under ultrasound guidance on early motor function after total knee arthroplasty. Braz J Anesthesiol. 2022 Jan-Feb;72(1):110-114. doi: 10.1016/j.bjane.2021.04.012. Epub 2021 Apr 26. PMID 33915199
- [Background] Nobre LV, Cunha GP, Sousa PCCB, Takeda A, Cunha Ferraro LH. [Peripheral nerve block and rebound pain: literature review]. Braz J Anesthesiol. 2019 Nov-Dec;69(6):587-593. doi: 10.1016/j.bjan.2019.05.001. Epub 2019 Nov 2. PMID 31690509
- [Background] Admassie BM, Tegegne BA, Alemu WM, Getahun AB. Magnitude and severity of rebound pain after resolution of peripheral nerve block and associated factors among patients undergoes surgery at university of gondar comprehensive specialized hospital northwest, Ethiopia, 2022. Longitudinal cross-sectional study. Ann Med Surg (Lond). 2022 Nov 18;84:104915. doi: 10.1016/j.amsu.2022.104915. eCollection 2022 Dec. PMID 36536717
- [Background] Lavand'homme P. Rebound pain after regional anesthesia in the ambulatory patient. Curr Opin Anaesthesiol. 2018 Dec;31(6):679-684. doi: 10.1097/ACO.0000000000000651. PMID 30124544
- [Background] Williams BA, Bottegal MT, Kentor ML, Irrgang JJ, Williams JP. Rebound pain scores as a function of femoral nerve block duration after anterior cruciate ligament reconstruction: retrospective analysis of a prospective, randomized clinical trial. Reg Anesth Pain Med. 2007 May-Jun;32(3):186-92. doi: 10.1016/j.rapm.2006.10.011. PMID 17543812
- [Background] Munoz-Leyva F, Cubillos J, Chin KJ. Managing rebound pain after regional anesthesia. Korean J Anesthesiol. 2020 Oct;73(5):372-383. doi: 10.4097/kja.20436. Epub 2020 Aug 10. PMID 32773724
- [Background] Hade AD, Okano S, Pelecanos A, Chin A. Factors associated with low levels of patient satisfaction following peripheral nerve block. Anaesth Intensive Care. 2021 Mar;49(2):125-132. doi: 10.1177/0310057X20972404. Epub 2021 Mar 30. PMID 33784851
- [Background] Dada O, Gonzalez Zacarias A, Ongaigui C, Echeverria-Villalobos M, Kushelev M, Bergese SD, Moran K. Does Rebound Pain after Peripheral Nerve Block for Orthopedic Surgery Impact Postoperative Analgesia and Opioid Consumption? A Narrative Review. Int J Environ Res Public Health. 2019 Sep 5;16(18):3257. doi: 10.3390/ijerph16183257. PMID 31491863
- [Background] Barry GS, Bailey JG, Sardinha J, Brousseau P, Uppal V. Factors associated with rebound pain after peripheral nerve block for ambulatory surgery. Br J Anaesth. 2021 Apr;126(4):862-871. doi: 10.1016/j.bja.2020.10.035. Epub 2020 Dec 31. PMID 33390261
- [Background] Fang J, Shi Y, Du F, Xue Z, Cang J, Miao C, Zhang X. The effect of perineural dexamethasone on rebound pain after ropivacaine single-injection nerve block: a randomized controlled trial. BMC Anesthesiol. 2021 Feb 12;21(1):47. doi: 10.1186/s12871-021-01267-z. PMID 33579199
- [Background] Abrisham SM, Ghahramani R, Heiranizadeh N, Kermani-Alghoraishi M, Ayatollahi V, Pahlavanhosseini H. Reduced morphine consumption and pain severity with transdermal fentanyl patches following total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2014 Jul;22(7):1580-4. doi: 10.1007/s00167-012-2287-9. Epub 2012 Dec 2. PMID 23212185
- [Background] van Bastelaere M, Rolly G, Abdullah NM. Postoperative analgesia and plasma levels after transdermal fentanyl for orthopedic surgery: double-blind comparison with placebo. J Clin Anesth. 1995 Feb;7(1):26-30. doi: 10.1016/0952-8180(94)00000-t. PMID 7772354
- [Background] Minville V, Lubrano V, Bounes V, Pianezza A, Rabinowitz A, Gris C, Samii K, Fourcade O. Postoperative analgesia after total hip arthroplasty: patient-controlled analgesia versus transdermal fentanyl patch. J Clin Anesth. 2008 Jun;20(4):280-3. doi: 10.1016/j.jclinane.2007.12.013. PMID 18617126
- [Background] Nelson L, Schwaner R. Transdermal fentanyl: pharmacology and toxicology. J Med Toxicol. 2009 Dec;5(4):230-41. doi: 10.1007/BF03178274. PMID 19876859
- [Background] Grond S, Radbruch L, Lehmann KA. Clinical pharmacokinetics of transdermal opioids: focus on transdermal fentanyl. Clin Pharmacokinet. 2000 Jan;38(1):59-89. doi: 10.2165/00003088-200038010-00004. PMID 10668859
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134